CLINICAL TRIAL: NCT00767572
Title: Effects of Statins on Endothelial Function in Patients With Coarctation of the Aorta
Brief Title: Statins and Endothelial Function in Patients With Coarctation of the Aorta
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H7151-32792-01
Record Dates: First submitted 2008-09-24; First posted 2008-10-07 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Coarctation of the Aorta
Keywords: Coarctation of the aorta; cross over design; atorvastatin; endothelial function
MeSH Terms: conditions — Aortic Coarctation | interventions — Atorvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin (Experimental): Patients are randomized to either atorvastatin or placebo once daily for 12 weeks. There is a 4 week washout, and then the groups are switched for 12 weeks. Brachial artery assessment will be performed before and after each 12 week period on therapy.
  Interventions: Drug: atorvastatin
- sugar pill (Placebo Comparator): See above. Patients will be randomized to atorvastatin vs. placebo for 12 weeks and after a 4 week washout period the groups will be switched.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin 80mg daily vs. placebo daily X 12 weeks, then 4 week washout period, then cross over groups to complete another 12 weeks. (Total study time is 28 weeks (12+4+12)
  Other Names: Lipitor
  Arms: atorvastatin
Drug: Sugar pill — atorvastatin 80mg daily vs. placebo daily X 12 weeks, then 4 week washout, then cross over groups X 12 weeks. Total study time is 28weeks (12+4+12).
  Other Names: placebo
  Arms: sugar pill

SUMMARY:
Coarctation of the aorta (CoA) accounts for approximately 8% of all congenital heart problems. Patients with CoA are well known to have an increased rates of early heart disease, high blood pressure, heart failure and stroke. Abnormal arterial function (dilation and constriction of the blood vessels) has been observed in these patients and likely contributes to the increased risk of cardiovascular problems. However, therapies targeted at improving arterial function have not been investigated in this population. Statin therapy (cholesterol medicines like Lipitor) have been studied in other subgroups of patients with abnormal arterial function and has shown benefit in improving arterial function and reducing risk of cardiovascular problems.

The investigators hypothesize that patients with CoA have abnormal arterial function leading to increased cardiovascular risk. We further hypothesize that statin therapy may improve this problem. We plan to compile a complete database of information regarding these patients cardiovascular health and propose to then examine the effect of atorvastatin (Lipitor) on arterial function as measured by changes in arm arterial function tests.

DETAILED DESCRIPTION:
The study design is a randomized double-blind cross over clinical trial. Patients who meet inclusion criteria and no exclusion criteria will be enrolled. They will undergo a baseline cardiovascular assessment including echocardiography, magnetic resonance imaging or magnetic resonance angiography (MRI/MRA), serum blood samples, brachial artery reactivity testing, and carotid intimal media thickness testing. Once they have completed their baseline testing, they will be randomized to either atorvastatin 80mg or placebo. They will complete 12 weeks of therapy and return at the end of 12 weeks to have a repeat brachial artery study and serum studies. There will then be a four week washout period where they take no medication. They will return for a follow up visit at the end of that four week period for repeat baseline brachial artery testing and serum studies. They then will be assigned to the opposite agent they were on previously (so if they originally were on placebo they switch to atorvastatin and vice versa). They will complete another 12 weeks of therapy and return at the end for a final brachial artery study and blood testing.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18 years with repaired coarctation of the aorta (CoA) and willing to participate in all portions of the study including follow up, blood draws, urine sample, echocardiogram, MRI, brachial artery flow-mediated dilatation (FMD) testing, Carotid Intima Media Thickness (CIMT) testing and statin administration.

Exclusion Criteria:

* patients who are pregnant, nursing, or planning on becoming pregnant in the subsequent year
* current smokers
* patients with documented coronary artery disease (CAD), other systemic inflammatory disorder such as systemic lupus erythematosis or rheumatoid arthritis
* patients already on statin therapy or who have had previous adverse effects to statin therapy
* patients with hepatic transaminases >2X the upper limit of normal
* patients with creatinine clearance <60mg/dL
* patients who have implanted devices such as pacemakers or defibrillators that preclude MRI testing
* patients with low blood pressure at baseline (< 90/50)
* patients who are unwilling or unable to comply with the aforementioned portions of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Medical Center, 505 Parnassus Ave, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the UCSF Adult Congenital Heart Disease Clinic between July 2008 and July 2009. All reviewed the study protocol and agreed to participate. There was no compensation for study participants.
Pre-assignment Details: Patients were excluded if they did not have prior repair of aortic coarctation or could not participate in all 4 study visits.
Groups:
- Atorvastatin Then Sugar Pill, or Sugar Pill Then Atorvastatin: Patients were randomized to atorvastatin or placebo once daily for 12 weeks. After a 4 week washout, each participant received the other intervention for 12 weeks. Brachial artery assessment was performed before and after each 12 week intervention.
Period: First Intervention (12 Weeks)
Arm/Group | Atorvastatin Then Sugar Pill, or Sugar Pill Then Atorvastatin
Started | 12
Completed | 12
Not Completed | 0
Period: Washout (4 Weeks)
Arm/Group | Atorvastatin Then Sugar Pill, or Sugar Pill Then Atorvastatin
Started | 12
Completed | 12
Not Completed | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Atorvastatin Then Sugar Pill, or Sugar Pill Then Atorvastatin
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin Then Sugar Pill, or Sugar Pill Then Atorvastatin: Patients were randomly assigned to receive atorvastatin or placebo once daily for 12 weeks. After a 4 week washout, each participant received the other intervention for 12 weeks. Brachial artery assessment were performed before and after each 12 week intervention.
Arm/Group | Atorvastatin Then Sugar Pill, or Sugar Pill Then Atorvastatin
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Pre-post Change in Brachial Artery Reactivity
Description: Brachial artery reactivity was assessed by Flow-mediated dilatation (FMD), performed before and after the 12 week period on therapy. FMD uses high-frequency ultrasound measurement of changes in brachial artery diameter after a 5-minute blood pressure cuff arterial occlusion. Brachial artery reactivity has been shown to predict long-term cardiovascular events.
Time Frame: Baseline, 12 weeks
Population: 12 enrolled participants were randomly assigned to receive a 12-week course of either atorvastatin or placebo, followed by a 4-week washout, then 12 weeks on the alternate intervention.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Atorvastatin: Patients are randomized to either atorvastatin or placebo once daily for 12 weeks. There is a 4 week washout, and then the groups are switched for 12 weeks.
Arm/Group | Atorvastatin | Sugar Pill
Number analyzed (Participants) | 12 | 12
mm | 3 (1.5) | 3 (1.5)
Statistical Analysis 1: Comparison: Atorvastatin vs Sugar Pill; Null hypothesis: pre-post brachial artery diameter changes do not differ between placebo and atorvastatin; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Significance threshold p<0.05

ADVERSE EVENTS:
Arm/Group | Atorvastatin | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
All patients were enrolled and completed the study interventions and assessments. Technical problems with measurements may have led to some unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No